CLINICAL TRIAL: NCT01238835
Title: Placement of AoRtic Balloon Expandable Transcatheter VAlves TrIaL (TransApical)
Brief Title: PREVAIL-TA: Placement of Aortic Balloon Expandable Transcatheter Valves Trial (Europe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-06
Record Dates: First submitted 2010-01-26; First posted 2010-11-11 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Sapien XT Valve; Valvular Heart Disease; Aortic Stenosis; Heart Valve Therapy; Transapical; Transcatheter
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVR-TA (Experimental): Transcatheter valve replacement with transapical access
  Interventions: Device: SAPIEN XT™ Transapical aortic valve replacement

INTERVENTIONS:
Device: SAPIEN XT™ Transapical aortic valve replacement — Transcatheter aortic valve implantation via the transapical approach
  Other Names: Sapien XT; Next generation Ascendra delivery system inclusive accessory

SUMMARY:
A single arm, prospective multicenter non-randomized confirmatory clinical trial evaluating the Edwards SAPIEN XT™ transcatheter heart valve (model 9300TFX; "study valve"), the next generation Ascendra™ transapical delivery system, and crimper accessories.

DETAILED DESCRIPTION:
Purpose: The purpose of this trial is to evaluate the acute safety and effectiveness of the SAPIEN XT™ study valve and next generation Ascendra™ delivery components.

Follow-up Intervals: Subject data collection will include clinical information at baseline and during the index procedure. Subjects will undergo clinical follow-up at discharge, 30 days, 6 month annually for 5 years.

ELIGIBILITY:
Inclusion:

1. EuroSCORE of ≥ 15 %
2. Severe senile degenerative aortic valve stenosis
3. Symptomatic aortic valve stenosis
4. Informed consent
5. Compliance

Exclusion:

1. Logistic Euroscore > 40 %
2. Evidence of an acute myocardial infarction
3. Congenital unicuspid or congenital bicuspid valve/ non-calcified
4. Mixed aortic valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Thomas Walther, Principal Investigator — Kerckhoff Klinik; Dr. Olaf Wendler, Principal Investigator — King's College London
Locations (20):
- Medizinische Universitat Wien Univ.Klinik f.Chirurgie, Vienna, Austria
- Hôspital Bichat, Paris, France
- Germany (16):
  - Herz-Und Gefasszentrum Bad Bevensen, Bad Bevensen
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz-und-Gefass Klinik, Bad Neustadt an der Saale
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen
  - Schüchtermann-Klinik, Bad Rothenfelde
  - Heart Center University Cologne, Cologne
  - Herzzentrum Dresden GmbH, Dresden
  - University Clinic Erlangen, Erlangen
  - University Hospital Essen, West German Heart Center, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Cardiac Surgery Karlsruhe, Karlsruhe
  - Heart Center Leipzig, Leipzig
  - German Heart Center Munich, Munich
  - University Hospital Munich-Grosshadern, Munich
  - Hospital Munich-Bogenhausen, Munich
  - Robert-Bosch-Krankenhaus, Stuttgart
- United Kingdom (2):
  - St. Thomas' Hospital - NHS Trust, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One patient withdrew from the study prior to procedure and one patient did not continue to procedure due to poor health.
Pre-assignment Details: Two enrolled subjects did not enter the procedure room.
Period: Overall Study
Arm/Group | TAVR-TA
Started | 218
Completed | 82
Not Completed | 136
Not completed — Death | 124
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 1
Not completed — Site early discontinuation | 2

BASELINE CHARACTERISTICS:
Population: As treated population
Arm/Group | TAVR-TA
Number analyzed (Participants) | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.2 (5.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 153
Logistic EuroSCORE [Mean (Standard Deviation); unit: Units on a scale] — The logistic European System for Cardiac Operative Risk Evaluation (logistic EuroSCORE) measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk of operative mortality.
  Units on a scale | 24.0 (7.27)
NYHA Class [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV. I = no limitations of physical activity; II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath.; IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
  Participants
    Class I/II | 36
    Class III/IV | 182

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths
Description: Number of death at 30-days from the index procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR-TA
Number analyzed (Participants) | 218
Participants | 16

2. Secondary Outcome: Number of Participants With a Stroke
Description: Total Number of Participants with a Stroke.
Time Frame: 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | TAVR-TA
Number analyzed (Participants) | 218
Participants | 4

ADVERSE EVENTS:
Time Frame: 5 Years
Description: All adverse events are site reported
Arm/Group | TAVR-TA
All-Cause Mortality (participants affected / at risk) | 124/218
Serious Adverse Events (participants affected / at risk) | 201/218
Other Adverse Events (participants affected / at risk) | 212/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR-TA (N=218)
Access Related Complication - Thoracic (Injury, poisoning and procedural complications) | 3 (3)
Access Related Complication - Ventricle (Injury, poisoning and procedural complications) | 3 (3)
Aneurysm (Vascular disorders) | 2 (2)
Angina (Cardiac disorders) | 10 (10)
Annular Dissection (Injury, poisoning and procedural complications) | 1 (1)
Arrhythmia Supraventricular (Cardiac disorders) | 15 (19)
Arrhythmia Ventricular (Cardiac disorders) | 7 (8)
Bleeding - Not Trauma Not Procedure (Vascular disorders) | 10 (10)
Bleeding - Procedure (Injury, poisoning and procedural complications) | 13 (17)
Bleeding - Trauma (Injury, poisoning and procedural complications) | 5 (5)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (24)
Coagulopathy / Hematological Disorder (Blood and lymphatic system disorders) | 53 (68)
Conduction Defects w/o Permanent Pacemaker (Cardiac disorders) | 1 (1)
Conduction Defects with Permanent Pacemaker (Cardiac disorders) | 32 (35)
Decubitus (Skin and subcutaneous tissue disorders) | 1 (1)
Delivery System Malfunction (Product Issues) | 1 (1)
Drug Reaction (General disorders) | 1 (1)
Endocarditis (Infections and infestations) | 7 (8)
Gastro-Intestinal Event (Gastrointestinal disorders) | 29 (39)
Heart Failure (Cardiac disorders) | 58 (90)
Hemodynamic Collapse (Vascular disorders) | 17 (18)
Hypertension (Vascular disorders) | 7 (10)
Hypotension (Vascular disorders) | 3 (3)
Infection / Inflammation (Infections and infestations) | 62 (90)
Metabolic Disorder (Metabolism and nutrition disorders) | 5 (5)
Mitral Regurg. ( 3+ or 4+) (Cardiac disorders) | 2 (2)
Mitral Valve Compromise (Injury, poisoning and procedural complications) | 1 (1)
Multiple Organ Failure (General disorders) | 8 (8)
Myocardial Infarction (Cardiac disorders) | 10 (14)
Neurological Event Minor - Not Stroke (Nervous system disorders) | 9 (13)
Neurological Event Severe - Not Stroke (Nervous system disorders) | 9 (10)
Non-Struct Valve Dysf. (Not PVL) (General disorders) | 1 (1)
Orthopedic Event (General disorders) | 17 (23)
Other (General disorders) | 67 (114)
Perivalvular Leak (1+ or 2+) (Product Issues) | 1 (1)
Perivalvular Leak (3+ or 4+) (Product Issues) | 7 (7)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 28 (31)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure requiring Permanent Dialysis (>30d) (Renal and urinary disorders) | 2 (2)
Renal Insufficency not requiring Dialysis (Renal and urinary disorders) | 17 (20)
Renal Insufficiency / Failure requiring Temporary Dialysis (< or = 30d) (Renal and urinary disorders) | 19 (21)
Respiratory Comp / Failure not requ. Resp Assistance (Respiratory, thoracic and mediastinal disorders) | 17 (19)
Respiratory Comp / Failure requ. Resp Assistance (Respiratory, thoracic and mediastinal disorders) | 25 (31)
Sepsis (Infections and infestations) | 17 (19)
Stroke - Embolic / Ischemic Origin (Nervous system disorders) | 12 (12)
Stroke - Unknown Origin (Nervous system disorders) | 3 (3)
Struct Valve Deterioration (SVD) (Injury, poisoning and procedural complications) | 1 (1)
Sudden Death (General disorders) | 20 (20)
Syncope (Nervous system disorders) | 7 (9)
Thoracic Wound Comp. (Injury, poisoning and procedural complications) | 6 (8)
Thrombus (Vascular disorders) | 1 (1)
Transitory Psychotic Syndrome (Psychiatric disorders) | 9 (9)
Valve Embolization (General disorders) | 1 (1)
Vascular Event (Not Access-Related) (Vascular disorders) | 17 (27)
Ventricular / Myocardial Injury / Perforation (Injury, poisoning and procedural complications) | 1 (1)
Vision Disorder (Eye disorders) | 3 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR-TA (N=218)
Arrhythmia Supraventricular (Cardiac disorders) | 64 (75)
Bleeding - Procedure (Injury, poisoning and procedural complications) | 12 (12)
Coagulopathy / Hematological Disorder (Blood and lymphatic system disorders) | 34 (38)
Conduction Defects w/o Permanent Pacemaker (Cardiac disorders) | 17 (18)
Gastro-Intestinal Event (Gastrointestinal disorders) | 36 (49)
Heart Failure (Cardiac disorders) | 23 (27)
Hypertension (Vascular disorders) | 15 (16)
Infection / Inflammation (Infections and infestations) | 94 (142)
Metabolic Disorder (Metabolism and nutrition disorders) | 27 (31)
Neurological Event Minor - Not Stroke (Nervous system disorders) | 26 (29)
Orthopedic Event (General disorders) | 16 (17)
Other (General disorders) | 122 (253)
Pericardial Effusion (Cardiac disorders) | 13 (14)
Peripheral Edema (General disorders) | 30 (34)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 130 (143)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 18 (18)
Renal Insufficency not requiring Dialysis (Renal and urinary disorders) | 36 (39)
Respiratory Comp / Failure not requ. Resp Assistance (Respiratory, thoracic and mediastinal disorders) | 25 (32)
Transitory Psychotic Syndrome (Psychiatric disorders) | 39 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes